CLINICAL TRIAL: NCT00865241
Title: A Relative Bioavailability Study of 5 mg Glyburide/500 mg Metformin HCl Tablets Under Fasting Conditions
Brief Title: A Relative Bioavailability Study of Glyburide/Metformin HCl 5 mg/500 mg Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Meena Venugopal, Director, Clinical R&D, Actavis Inc
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: R02-994
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Metformin; Glyburide; Healthy subjects
MeSH Terms: interventions — Glyburide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Glyburide and Metformin Hydrochloride Tablets 5 mg/500 mg, single dose
  Interventions: Drug: Glyburide and Metformin Hydrochloride Tablets 5 mg/500 mg
- B (Active Comparator): CLUCOVANCE® 5 mg/500 mg Tablets, single dose
  Interventions: Drug: CLUCOVANCE® 5 mg/500 mg Tablets, single dose

INTERVENTIONS:
Drug: Glyburide and Metformin Hydrochloride Tablets 5 mg/500 mg — A: Experimental Subjects received Alpharma formulated products under fasting conditions
  Other Names: Glyburide; Metformin
  Arms: A
Drug: CLUCOVANCE® 5 mg/500 mg Tablets, single dose — B: Active comparator Subjects received Bristol-Myers Squibb Company formulated products under fasting conditions
  Other Names: Glyburide; Metformin
  Arms: B

SUMMARY:
The purpose of this study is to compare the relative bioavailability of 5 mg Glyburide/500 mg Metformin Hydrochloride Tablets by Purepac Pharmaceutical Co. with that of 5 mg/500 mg CLUCOVANCE® Tablets by Bristol-Myers Squibb Company following a single oral dose (1 x 5 mg/500 mg tablet) in healthy adult volunteers under fasting conditions.

DETAILED DESCRIPTION:
Study Type: Interventional Study Design: Randomized, single dose, two way crossover study under fasting conditions

Official Title: A Relative Bioavailability Study of 5 mg Glyburide/500 mg Metformin HCl Tablets Under Fasting Conditions

Further study details as provided by Actavis Elizabeth LLC:

Primary Outcome Measures:

Rate and Extend of Absorption

ELIGIBILITY:
Inclusion Criteria:

1. Screening Demographics: All volunteers selected for this study will be healthy men or women 18 years of age or older at the time of dosing. The weight range will not exceed ± 20% for height and body frame as per Desirable Weights for Adults -1983 Metropolitan Height and Weight Table.
2. Screening Procedures: Each volunteer will complete the screening process within 28 days prior to Period I dosing. Consent documents for both the screening evaluation and HIV antibody determination will be reviewed, discussed, and signed by each potential participant before full implementation of screening procedures.

   Screening will include general observations, physical examination, demographics, medical and medication history, an electrocardiogram, sitting blood pressure and heart rate, respiratory rate and temperature. -The physical examination will include, but may not be limited to, an evaluation of the cardiovascular, gastrointestinal, respiratory and central nervous systems.

   The screening clinical laboratory procedures will include:
   * HEMATOLOGY: hematocrit, hemoglobin, WBC count with differential; RBC count, platelet count;
   * CLINICAL CHEMISTRY: serum creatinine, BUN, glucose, AST(GOT), ALT(GPT), albumin, total bilirubin, total protein, and alkaline phosphatase;
   * HIV antibody and hepatitis B surface antigen screens;
   * URINALYSIS: by dipstick, microscopic examination if dipstick positive; and .
   * URINE DRUG SCREEN: ethyl alcohol, amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine metabolites, opiates and phencyclidine.
   * SERUM PREGNANCY SCREEN (female volunteers only)
3. If female and:

   * of childbearing potential, is practicing an acceptable barrier method of birth control for the duration of the study as judged by the investigator(s), such as condoms, sponge, foams, jellies, diaphragm; intrauterine device (IUD), or abstinence; or
   * is postmenopausal for at least I year; or
   * is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).

Exclusion Criteria:

1. Volunteers with a recent history of drug or alcohol addiction or abuse.
2. Volunteers with the presence of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease (as determined by the medical investigator).
3. Volunteers whose clinical laboratory test values are outside the accepted reference range and when confirmed on re-examination are deemed to be clinically significant.
4. Volunteers demonstrating a positive hepatitis B surface antigen screen or a reactive HIV antibody screen.
5. Volunteers demonstrating a positive drug abuse screen when screened for this study.
6. Female volunteers demonstrating a positive pregnancy screen.
7. Female volunteers who are currently breastfeeding.
8. Volunteers with a history of allergic response(s) to glyburide, metformin or related drugs.
9. Volunteers with a history of clinically significant allergies including drug allergies.
10. Volunteers with a clinically significant illness during the 4 weeks prior to Period I dosing (as determined by the medical investigator).
11. Volunteers who currently use tobacco products.
12. Volunteers who have taken any drug known to induce or inhibit hepatic• drug metabolism in the 28 days prior to Period I dosing.
13. Volunteers who report donating greater than 150 mL of blood within 28 days prior to Period I dosing. All subjects will be advised not to donate blood for four weeks after completing the study.
14. Volunteers who have donated plasma (e.g. plasmapheresis) within 14 days prior to Period I dosing. All subjects will be advised not to donate plasma for four weeks after completing the study.
15. Volunteers who report receiving any investigational drug within 28 days prior to Period I dosing.
16. Volunteers who report taking any systemic prescription medication in the 14 days prior to Period I dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2002-11; Primary Completion 2002-11 (Actual); Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Rate and Extend of Absorption | 36 hours

CONTACTS AND LOCATIONS:
Overall Officials: James D. Carlson,, Pharm.D,, Principal Investigator — PRACS Institute, Ltd.
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States